CLINICAL TRIAL: NCT04496973
Title: University of Delaware Participant Recruitment Registry for Parkinson's Disease Research
Brief Title: University of Delaware Parkinson's Disease Registry
Status: Recruiting | Type: Observational
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Roxana Burciu, Roxana Burciu, PhD, University of Delaware
Other Study IDs: 1535874
Record Dates: First submitted 2020-07-29; First posted 2020-08-04 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this Parkinson's Disease Registry is to assist with recruitment of willing participants into future Parkinson's disease research studies at the University of Delaware.

DETAILED DESCRIPTION:
There is an urgent need for Parkinson's Disease research due to its increasing global prevalence. Participant recruitment is a significant challenge to the success of Parkinson's disease research and we need your help more than ever in moving the field forward and improving the lives of people who have Parkinson's disease. Recruitment of study participants can be facilitated by maintaining registries of people who agree to be contacted for future studies.

The purpose of the University of Delaware Participant Recruitment Registry for Parkinson's Disease Research is to create a registry that includes the contact information and basic health information pertaining the participant's diagnosis of Parkinson's disease. The registry will streamline recruitment and enrollment in a variety of research studies focusing on topics such as, but not limited to: brain changes in Parkinson's disease, balance and gait in Parkinson's disease, exercise and its effect on motor function.

To be in the registry individuals must have a clinical diagnosis of Parkinson's Disease and have an interest in participating in research studies.

To become a member of this registry, primary information including contact information and some general medical information are needed.

ELIGIBILITY:
Inclusion Criteria:

* Individual 21 years old or older
* A clinical diagnosis of Parkinson's disease
* Interest in participating in one or more investigator-led research studies at the University of Delaware

Exclusion Criteria:

* Individuals with a clinical diagnosis of parkinsonism that is not considered primary (e.g. vascular parkinsonism) or an atypical parkinsonian syndrome (e.g., progressive supranuclear palsy, multiple system atrophy, corticobasal degeneration etc.)
* Clinical diagnosis of dementia

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who have a clinical diagnosis of Parkinson's disease and are interested in participating in Parkinson's disease research studies University of Delaware.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-05-28 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Parkinson's Disease Diagnosis | Once a year, at the beginning of the year
  By following up once a year, we will evaluate a participant's medical history to validate a diagnosis of Parkinson's Disease. A confirmed diagnosis of Parkinson's Disease is a criteria for continuing to be a part of the registry.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No